CLINICAL TRIAL: NCT07055932
Title: Effectiveness of an Interactive School-Based Oral Health Education Program in Reducing Periodontal Disease Among Palestinian Adolescents: A Double-Blinded Intervention Study
Brief Title: Interactive School-Based Oral Health Education Program to Reduce Periodontal Disease in Palestinian Adolescents
Acronym: ISBOHE-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Quds University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REF.13/24
Record Dates: First submitted 2025-06-12; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-05

CONDITIONS: Periodontal Diseases
Keywords: interactive school-based education
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: In this parallel-assignment design, eligible ninth-grade students are randomized by school into either the interactive oral health education arm (intervention group) or the standard lecture arm (one educational session) (control group). Each participant remains in their assigned group for the full two-month intervention period, with no crossover between arms. Outcomes are assessed at baseline and two months post-intervention to compare changes in periodontal and oral hygiene indices and oral hygiene, dietary, and smoking behaviors between the two fixed groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding was applied at the participant and outcome assessor levels. Participants were not informed of their group allocation, and assessors conducting data collection were blinded to reduce assessment bias. The educator administering the intervention was not blinded, as this was not operationally feasible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Interactive Oral Health Education (Experimental): Participants in this arm receive an interactive oral health education program consisting of six sessions delivered over two months (one session every 10 days). Each session lasts 30-45 minutes and includes interactive lectures, visual presentations (PowerPoint slides and photographs), and anatomical models (tooth and gum replicas). Practical components involve live demonstrations of cleaning techniques (tooth brushing and flossing), group discussions, and educational puzzles. The aim is to strengthen participants' knowledge and hands-on practice of oral and periodontal hygiene habits, as well as to raise awareness of risks related to smoking and dietary factors.
  Interventions: Behavioral: "Interactive Oral Health Education Program"
- Control Group - Single Oral Hygiene Session (No Intervention): Participants in this arm receive a single oral hygiene session at the beginning of the study. This session provides a straightforward explanation of tooth brushing and flossing techniques, without any additional interactive components or ongoing follow-up. The purpose is to measure improvements resulting from the interactive education compared to one-time standard care.

INTERVENTIONS:
Behavioral: "Interactive Oral Health Education Program" — The interactive program in this study is distinguished by its multi-modal, hands-on approach and its sustained, bi-weekly delivery over two months, whereas most other school-based interventions rely on a single lecture or short-term animation. Specifically, our program:
  Combines interactive lectures with live demonstrations (brushing/flossing on models), group discussions, and educational puzzles to reinforce learning through active participation rather than passive listening.
  Uses anatomical tooth-and-gum replicas alongside PowerPoint slides and photographs to bridge theory and practice within each 30-45-minute session.
  Addresses periodontal risk factors (e.g., smoking, diet) in dedicated sessions, integrating behavioural change techniques (e.g., problem-solving brainstorming, personalized feedback) rather than focusing solely on plaque removal.
  Is delivered in six sessions (one every 10 days) to maximize retention and allow for iterative skill practice, unlike brief "brush-along"
  Arms: Intervention Group - Interactive Oral Health Education

SUMMARY:
The goal of this intervention study was to evaluate the effectiveness of a two-month interactive school-based oral health education program in reducing periodontal disease and improving oral health behaviors among 15-year-old schoolchildren in Nablus, Palestine.

The study was guided by the following hypotheses:

* The interactive education program would lead to a significant reduction in Community Periodontal Index for Treatment Needs (CPITN) and Simplified Oral Hygiene Index (S-OHI) scores.
* The program would result in significant improvements in oral hygiene practices, dietary habits, and smoking behaviors compared to standard oral health education.

Researchers compared students who received six interactive oral health sessions over two months to those who received a single standard oral health lecture, to determine whether the intervention group experienced greater improvements in periodontal status and self-reported health behaviors.

Participants:

* Completed self-administered questionnaire assessing oral hygiene practices, dietary habits, and smoking behaviors
* Underwent clinical periodontal examinations using CPITN and S-OHI indices
* Participated in oral health education sessions (intervention group only)

DETAILED DESCRIPTION:
This completed clinical trial evaluated the effectiveness of an interactive, school-based oral health education program in improving periodontal health and associated behaviors among 9th-grade students in Nablus City, Palestine. The study employed a double-blind, pre-test/post-test experimental design involving 946 students (536 intervention, 410 control) from 15 schools selected through stratified random sampling.

Baseline data collection occurred in March 2024 and included clinical assessments using the Community Periodontal Index for Treatment Needs (CPITN) and Simplified Oral Hygiene Index (S-OHI), along with a validated 47-item questionnaire measuring oral hygiene practices, dietary habits, and smoking behaviors. Following randomization by school, the intervention group received six interactive oral health education sessions, while the control group attended one standard lecture. Follow-up assessments took place two months later.

Two levels of blinding were implemented: participants were unaware of group assignment, and outcome assessors were blinded during clinical evaluations. The educational program combined audiovisual materials, live demonstrations, group discussions, and hands-on practice focused on oral anatomy, prevention and treatment of periodontal disease, smoking harms, and nutrition.

Primary outcomes included changes in CPITN and S-OHI scores. Secondary outcomes addressed self-reported improvements in oral hygiene, dietary behaviors, and smoking habits. Data analysis was performed using SPSS version 25.0, with paired and independent t-tests applied to evaluate within- and between-group differences.

The findings indicated significant improvements in the intervention group across all primary and secondary outcomes. These results support the program's effectiveness in enhancing periodontal health and related behaviors among adolescents through interactive, school-based education.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents enrolled in 9th grade at one of the selected governmental or private schools in Nablus City during the 2023-2024 academic year
* Age approximately 15 years (index age for adolescence as defined by the World Health Organization)
* Willingness to participate and availability for both baseline and two-month follow-up assessments
* Provision of written informed consent by a parent or legal guardian, and written assent by the student
* Ability to complete the study questionnaire and undergo clinical periodontal and oral hygiene examinations

Exclusion Criteria:

* Students who were absent from school for medical or other reasons at the time of baseline screening
* Inability or unwillingness to comply with study procedures (e.g., not completing the questionnaire, refusing periodontal examination)
* Refusal to provide either parental/guardian consent or student assent

Ages: 15 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 946 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Mean Community Periodontal Index of Treatment Needs (CPITN) Score | Baseline (prior to intervention) and two months post-intervention
  Change in Mean Community Periodontal Index of Treatment Needs (CPITN) Score The outcome is defined as the mean difference in the Community Periodontal Index of Treatment Needs (CPITN) score between baseline and two months post-intervention. The CPITN is a standardised index developed by the World Health Organisation to assess periodontal status. Scores were recorded using a WHO periodontal probe across six index teeth (teeth 16, 11, 26, 36, 31, and 46), and the mean score per participant was calculated.
  The Community Periodontal Index of Treatment Needs scale ranges from 0 to 4, where:
  * 0 = Healthy gingiva
  * 1 = Bleeding on probing
  * 2 = Presence of calculus
  * 3 = Shallow periodontal pockets (4-5 mm)
  * 4 = Deep periodontal pockets (6 mm or more) Higher scores indicate worse periodontal health.

SECONDARY OUTCOMES:
Mean Difference in Simplified Oral Hygiene Index (S-OHI) Score Pre- and Post-Intervention | From baseline (March 2024) to two months post-intervention (May 2024)
  Change in Mean Simplified Oral Hygiene Index (S-OHI) Score The outcome is defined as the mean difference in the Simplified Oral Hygiene Index (S-OHI) score between baseline and two months post-intervention. The S-OHI is a standardized tool developed by Greene and Vermillion to assess oral hygiene status through the presence of debris and calculus on specific index teeth (11, 16, 26, 31, 36, and 46).
  Each tooth surface was scored separately for debris and calculus, using a scale from 0 to 3 for each component. These scores were combined and averaged across examined surfaces to yield a final index score per participant.
  The total S-OHI score ranges from 0 to 6, where:
  * 0 = no debris
  * 1= debris on one-third of the tooth surface
  * 2=debris on two-thirds of the tooth surface
  * 3=debris on the all-tooth surface
Change in Mean Oral Hygiene Practices Score from Baseline to Two Months Post-Intervention | Baseline (March 2024) and 2 months post-intervention (May 2024)
  This outcome measures the change in oral hygiene practices using a composite score derived from questionnaire responses. Items assessed included brushing frequency, duration, technique, toothbrush type, and replacement frequency. Each item was scored on a scale from 0 to 3. Higher scores indicate more frequent and correct practices. The outcome is calculated as the mean difference between baseline and two months post-intervention.
Change in Mean Dietary Habits Score from Baseline to Two Months Post-Intervention | Baseline (March 2024) and two months post-intervention (May 2024)
  This outcome evaluates changes in dietary habits using a questionnaire-based composite score. Items covered breakfast frequency and intake of nutritious versus non-nutritious foods. Responses were coded into a continuous diet score, with higher scores reflecting healthier eating patterns. The outcome is defined as the mean difference between baseline and two months post-intervention.
Change in Mean Smoking Behaviors Score from Baseline to Two Months Post-Intervention | Baseline (March 2024) and two months post-intervention (May 2024)
  This outcome assesses changes in smoking-related behavior through a composite score. Questionnaire items included cigarette smoking frequency (times/week), number of cigarettes per day, and water-pipe use frequency. Responses were recoded so that higher scores reflect healthier behaviors (i.e., less frequent or no smoking). The mean score difference was calculated between baseline and post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Public Health, Al-Quds University, Abū Dīs, Jerusalem Governorate, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data (IPD) that underlie the results reported in this interventional study (including demographic variables, clinical measurements, and outcome assessments) will be made available beginning one year after publication for researchers who provide a methodologically sound proposal. Data will be shared via a public repository (e.g., Dryad) with a digital object identifier (DOI) to ensure persistent access. Interested investigators should contact the corresponding author (sura.kazlak@yahoo.com) to request data and submit a brief research proposal. Data will be provided under a data-use agreement prohibiting participants' re-identification and further sharing without permission.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be released 12 months after publication of results and remain available for 5 years thereafter.

REFERENCES:
- See also: Rice R. (2009). The effectiveness of computer-based interactive oral health education. MSc Thesis, Faculty of Medicine, University of Glasgow. Full text and appendices (e.g., questionnaires, intervention modules) available. — https://theses.gla.ac.uk/1017/
- Available data/document: Study Protocol — https://theses.gla.ac.uk/1017/

DOCUMENTS (3):
  • Study Protocol (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT07055932/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT07055932/SAP_001.pdf
  • Informed Consent Form (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT07055932/ICF_002.pdf